CLINICAL TRIAL: NCT02770573
Title: Long-term Response of Three Biomaterials Used as Desensitizer Agents Under Oral Environmental Exposure.
Brief Title: Use of Biomaterials as Desensitizer Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Egle Milia, Prof, Università degli Studi di Sassari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DH 2304/CE
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Dentin Sensitivity
Keywords: nano-hydroxyapatite
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with dentin hypersensitivity (Experimental): Patients with evident clinical signs of dentin hypersensitivity The following dental materials will be used following the manufacturers' instructions: Cavex Bite&White ExSense; Kuraray Teethmate™ Desensitizer; Ghimas Dentin Desensitizer.
  In view of the treatment with the desensitizing agents, teeth were randomly assigned into four groups.
  The application of the materials will be made only once. The effectiveness will be evaluated: immediately after application and after 1, 4, 12 weeks.
  Interventions: Other: Cavex Bite&White ExSense; Other: Kuraray Teethmate™ Desensitizer; Other: Ghimas Dentin Desensitizer

INTERVENTIONS:
Other: Cavex Bite&White ExSense — a water-based mint aroma gel containing hydroxyapatite and potassium nitrate.
Other: Kuraray Teethmate™ Desensitizer — Calcium-Phosphate-based powder and a liquid mainly water-based.
Other: Ghimas Dentin Desensitizer — a fluid desensitizing gel with 30% of nano-hydroxyapatite, added to 70:100 thousandths of micron-sized crystals of nano- hydroxyapatite.

SUMMARY:
Aim: to investigate the clinical effectiveness over 12 weeks of three different biomaterials, nano-hydroxyapatite based, in the therapy of the dental sensitivity.

Methods: The study is designed as a randomized clinical trial comparing: 1) Cavex Bite&White ExSense, 2) Teethmate™ Desensitizer , 3) Ghimas Dentin Desensitizer. The pain experience was generated by a cold stimulus directly to a sensitive tooth surface and assessed using the Visual Analogue Scale (VAS). The response was recorded before the application of the materials (PRE-1), immediately after (POST-1), at 1-week (POST-2), 4-weeks (POST-3) and 12-week controls (POST-4).

DETAILED DESCRIPTION:
Participants The study is designed as randomized clinical trial. The participants will be selected from the regular attenders of the Dental Clinic in the University of Sassari, Italy.

Inclusion criteria:

• patients will be considered suitable for the study if they have sensitive teeth showing abrasion, erosion, or recession with the exposure of the cervical dentine;

Exclusion criteria:

* teeth with subjective or objective evidence of carious lesions, pulpitis, restorations, premature contact, cracked enamel, active periapical infection, or which had received periodontal surgery or root-planning up to 6 months prior to the investigation will be excluded from the study
* professional desensitizing therapy during the previous 3 months, or use of desensitizing toothpaste in the last 6 weeks.
* Patients will be also excluded if they will be under significant medication that could interfere with pain perception (e.g., antidepressants, anti-inflammatory drugs, sedatives, and muscle relaxants).

Randomization Using a computer program (Excel 2010 for Mac OsX), the randomization will be carried on using an individual basis.

Clinical procedure A full medical and dental history will be taken and all the teeth will be carefully examined to confirm the diagnosis of DH. The experience of dentinal hypersensitivity and how this has affected the quality of life of the patients will be evaluated through a specific questionnaire. The nature and scope of the study will be explained and informed consent will be obtained.

A week before the experiment, patients received oral prophylaxis. Non-fluoride toothpaste, soft tooth- brush and oral hygiene instructions will be also provided in order to have standardized habits during the period of the study.

A week before the experiment, patients received oral prophylaxis. Non-fluoride toothpaste (Biorepair, Coswell), a soft toothbrush (Oral-B Sensitive Advantage, Procter & Gamble) and oral hygiene instructions were also provided. The level of sensitivity experienced by each patient was considered as independent of the position of the hypersensitive tooth in the oral cavity. The pain experience was assessed by a Visual Analogue Scale (VAS) using the methodology described in our previous study. The pain experience was measured using a VAS graded from 1 to 10. The pain stimulus was given by one examiner with the same equipment yielding similar air pressure each time, while another one performed the treatments.

Teeth will be randomly assigned to three groups (N= per group) for the treatment with the three desensitizing agents.

The following dental materials were used following the manufacturers' instructions:

1. Cavex Bite&White ExSense (Cavex Holland BV, RW Haarlem, The Netherlands), a water-based mint aroma gel containing hydroxyapatite and potassium nitrate.
2. Kuraray Teethmate™ Desensitizer (Kuraray Noritake Dental, Osaka, Japan), Calcium-Phosphate-based powder and a liquid mainly water-based.
3. Ghimas Dentin Desensitizer (Ghimas, Bologna, Italy), a fluid desensitizing gel with 30% of nano-hydroxyapatite, added to 70:100 thousandths of micron-sized crystals of nano- hydroxyapatite.

ELIGIBILITY:
Inclusion Criteria:

• patients will be considered suitable for the study if they had sensitive teeth showing abrasion, erosion, or recession with the exposure of the cervical dentine;

Exclusion Criteria:

* teeth with subjective or objective evidence of carious lesions, pulpitis, restorations, premature contact, cracked enamel, active periapical infection, or which had received periodontal surgery or root-planning up to 6 months prior to the investigation will be excluded from the study
* professional desensitizing therapy during the previous 3 months, or use of desensitizing toothpaste in the last 6 weeks.
* Patients will be also excluded if they will be under significant medication that could interfere with pain perception (e.g., antidepressants, anti-inflammatory drugs, sedatives, and muscle relaxants).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of change of dentinal hypersensitivity after treatment | before the treatment (PRE-1), immediately after (POST-1), after 1 week (POST-2), 4 weeks (POST-3), and 12 weeks (POST-4).
  The pain experience was assessed by a Visual Analogue Scale (VAS) using the methodology. The VAS scale consisted of a horizontal line that was 100 mm long, on which 'no pain' was marked on the right-hand extremity and 'unbearable pain' on the other. The patients expressed the intensity of the pain experienced by placing a mark at any point along the continuum. The distance, expressed in millimetres, from the right edge of 'no pain' was used as the VAS score. Each patient was asked to rate the perception of discomfort after the application of air via a dental syringe at 45-60 psi, 1 cm at the cervical third of the tooth after removing supragingival plaque with a low- speed handpiece with pumice powder and without fluoride. The adjacent teeth were covered by cotton rolls. The stimulus was delivered until reaction or up to a maximum duration of 10 s by the same examiner with the same equipment yielding similar air pressure each time.

CONTACTS AND LOCATIONS:
Overall Officials: Egle Milia, Prof, Principal Investigator — Università degli Studi di Sassari
Locations (1):
- Complex Operative Unit of Dentistry, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No
Not a plan for data sharing has been established. But, for anyone researcher would like to have this information, simply they may request them to us directly.

REFERENCES:
- [Background] Milia E, Castelli G, Bortone A, Sotgiu G, Manunta A, Pinna R, Gallina G. Short-term response of three resin-based materials as desensitizing agents under oral environmental exposure. Acta Odontol Scand. 2013 May-Jul;71(3-4):599-609. doi: 10.3109/00016357.2012.700063. Epub 2012 Aug 15. PMID 22891890
- [Background] Pinna R, Bortone A, Sotgiu G, Dore S, Usai P, Milia E. Clinical evaluation of the efficacy of one self-adhesive composite in dental hypersensitivity. Clin Oral Investig. 2015 Sep;19(7):1663-72. doi: 10.1007/s00784-014-1390-3. Epub 2015 Jan 23. PMID 25609032
- See also: Effectiveness of nano-hydroxyapatite toothpaste in reducing dentin hypersensitivity: a double-blind randomized controlled trial. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Derchi+G+Effectiveness+of+nano-hydroxyapatite+toothpaste+in+reducing+dentin+hypersensitivity%3A+A+double-blind+randomized+controlled+trial